CLINICAL TRIAL: NCT05581212
Title: Implementation of a New Strategic TB Case-Finding, Treatment and Prevention Public Health Pack in Thailand
Brief Title: TB Case-Finding, Treatment and Prevention Intervention in Thailand
Acronym: CaPThai
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Ministry of Health, Thailand (Other Government); London School of Hygiene and Tropical Medicine (Other); Tuberculosis and HIV Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRD-1-001; 21SANIN207 (Other Grant/Funding Number: Expertice France)
Record Dates: First submitted 2022-06-17; First posted 2022-10-14 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis
Keywords: Case-finding; Preventive treatment; Public Health Pack; Household contacts
MeSH Terms: conditions — Tuberculosis | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge Cluster Randomised Trial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Control phase) (No Intervention): In the current standard of care in Thailand, at time of diagnosis and tuberculosis (TB) treatment initiation, TB patients are being advised to tell their household (HH) contacts to consult at the TB clinic for screening and provision of either curative or preventive treatment - according to the screening outcome.
- Tuberculosis Case-Finding, Treatment and Prevention Public Health Pack (Intervention phase) (Experimental): In the selected provinces, individuals (≥18 years) with newly detected bacteriologically confirmed pulmonary Tuberculosis (index TB case) will be sensitized on the importance of HH contact investigation for detection and prevention of TB and stigma reduction.
  Index TB cases will be asked to enumerate all persons living in their HH for ≥1 month at the date of TB diagnostic (contact list), and provide their name/age/sex and relationship with the index case.
  Screening will be offered to each HH contact, using screening invitation cards that will be provided to the index TB case, to be handed over to each HH contact (or caregiver for children <13 years old).
  Urban and Village Health Volunteers (U/VHV),will visit the HH to enhance awareness of the importance of screening for TB case-finding and prevention and facilitate liaison with the hospital.
  If active tuberculosis has been formally excluded, they will be eligible to receive the Tuberculosis Preventive Treatment (TPT).
  Interventions: Other: Tuberculosis Case-Finding, Treatment and Prevention Public Health Pack

INTERVENTIONS:
Other: Tuberculosis Case-Finding, Treatment and Prevention Public Health Pack — Combined active case-finding, treatment and prevention of TB amongst HH contacts of TB cases, associated with initiation of standard of care (SOC) treatment in active TB cases and initiation of TB preventive therapy in those contacts without active TB, based on free screening. This intervention will be compared to the standard of care available in the country.
  Arms: Tuberculosis Case-Finding, Treatment and Prevention Public Health Pack (Intervention phase)

SUMMARY:
The project aimed to test a strategy for the early detection and prevention of tuberculosis in household contacts of tuberculosis patients in order to reduce the morbidity, mortality and transmission of this disease in Thailand. This strategy will be evaluated in comparison with the current programmatic approach through a pragmatic trial with cluster randomization (cluster randomized controlled trial) which will be conducted over the next 3 years. This project is carried out in collaboration with the Tuberculosis Division of the Ministry of Public Health of Thailand, the TB/HIV Research Foundation in Thailand and the London School of Hygiene and Tropical Medicine in England.

DETAILED DESCRIPTION:
Title: Implementation of a new Strategic TB Case-Finding, Treatment and Prevention Public Health Pack in Thailand (CapThai) Phase: IV, cluster randomized trial

Population:

adults (>= 18 years old) with pulmonary TB and their household contacts. Sites: 20 clusters (provincial hospitals) in Thailand

Duration of the study:

36 months

Subject participation duration:

9 months

Description of the intervention:

Combined active case-finding, treatment and prevention of TB amongst household contacts of TB cases, associated with initiation of SOC treatment in active TB cases and initiation of TB preventive therapy in those contacts without active TB, based on free screening. This intervention will be compared to the standard of care available in the country.

Overall objective:

To evaluate whether a public health intervention package focusing on the households of newly detected TB cases can increase active case-finding and uptake of TB preventive therapy in Thailand.

Specific objectives:

1. to compare the initiation and completion of TPT regimens amongst household contacts of infectious TB patients, overall and by gender and age group;
2. to evaluate the safety of short TPT regimens amongst HH contacts, overall and by gender and age group;
3. to compare the detection of TB and treatment uptake for active TB amongst HH contacts of infectious TB patients, overall and by gender and age group;
4. to assess the feasibility of the combined intervention among health care providers and beneficiaries, by gender and age group;
5. to assess the acceptability of the combined intervention among health care providers and beneficiaries, by gender and age group;
6. to evaluate the epidemiological impact of the combined intervention.

Study design:

The study uses a Stepped-Wedge Cluster Randomised Trial design. Randomisation will take place at the hospital level (cluster: provincial hospitals with >150 new TB cases/year). Twenty clusters will be enrolled and switch from the control to the intervention phase in four sequences every 3 months in a random order until all clusters are exposed to the intervention.

1. Intervention Phase: Newly detected bacteriologically confirmed TB patients (≥ 18 years) will be sensitized on the importance of HH contact investigation and TB stigma reduction. They will be asked to enumerate all contacts (name/age/sex/relationship) living in their HH for>1 month at the date of TB diagnostic. Screening invitation cards will be provided for each HH contact (or caregiver for children <13 years old), inviting them to attend the TB clinic at the selected hospital for free screening and evaluation. Transportation fees will be provided. Contacts detected with active TB will receive recommended treatment. In contacts for whom active TB is formally excluded, TPT will be initiated with the new short regimens: (i) children <2 years: isonicotine hydrazine (INH)+rifampicin daily for 3 months; (ii) children 2-12 years: INH+rifapentine weekly for 3 months; (iii) children≥13 and adults: INH+rifapentine daily for 1 month.
2. Control phase: current strategy relying on passive case detection and advice provided to TB patients to refer HH contacts to the TB clinic for screening. The index TB patient will be asked to enumerate HH contacts as above and inform them on the need to be screened at the TB clinic.

Endpoints:

Primary endpoint: Proportion of HH contacts with active TB excluded who are initiated on TPT within 4 weeks of the index TB patient diagnosis - overall, by age group (<15, ≥15 years) and gender.

Secondary endpoints:

1. Proportion of participants initiated on TPT who completed TPT;
2. Proportion of participants in the Intervention phase who were initiated on TPT for whom treatment is discontinued due to intolerance, adverse events, or severe adverse events;
3. Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 8 weeks of the index TB case diagnosis - overall, by age group (<15, ≥15 years) and gender;
4. Proportion of household contacts diagnosed with TB who completed TB treatment in the intervention vs. control phase;
5. Proportion of contacts receiving TPT who developed TB over the 9 months follow-up period in the intervention vs. control phase.

Estimated time to complete enrollment:

12-15 months

ELIGIBILITY:
Inclusion Criteria:

Inclusion of the index cases

* Age ≥18 years
* Newly bacteriologically confirmed TB case (within 1 month of diagnosis)
* Living in the same household for the last 3 months
* Reporting at least one HH contact
* Providing written informed consent for participation in the study

Inclusion of contacts

* All contacts living in the same HH, defined as any person who shared the same enclosed living space as the index TB case for one or more nights or for frequent or extended daytime periods for at least one month before the TB diagnosis is made.
* Providing written informed consent (signed by adult (≥18 years) contacts; or by parents/guardians for minors < 13 years or incapacitated people; written assent for children ≥13 years and < 18 years).

Exclusion Criteria:

Exclusion of index cases

* Index case who do not live in the catchment area of the study cluster
* Index cases diagnosed with rifampicin resistance, multidrug resistance (MDR) or extensively drug-resistant (XDR-TB)
* Index cases who are incarcerated

Exclusion of the contacts

- contact currently on TPT or on TB treatment or who finished such treatment in the last 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of household contacts with active tuberculosis excluded who are initiated on tuberculosis preventive treatment within 4 weeks of the index tuberculosis patient diagnosis - overall | Month18
  Proportion of household contacts with active tuberculosis excluded who are initiated on tuberculosis preventive treatment within 4 weeks of the index tuberculosis patient diagnosis - overall
Proportion of household contacts with active tuberculosis excluded who are initiated on tuberculosis preventive treatment within 4 weeks of the index tuberculosis patient diagnosis - by age group (<15, ≥15 years) | Month18
  Proportion of household contacts with active tuberculosis excluded who are initiated on tuberculosis preventive treatment within 4 weeks of the index tuberculosis patient diagnosis - by age group (<15, ≥15 years)
Proportion of household contacts with active tuberculosis excluded who are initiated on tuberculosis preventive treatment within 4 weeks of the index tuberculosis patient diagnosis - by gender | Month18
  Proportion of household contacts with active tuberculosis excluded who are initiated on tuberculosis preventive treatment within 4 weeks of the index tuberculosis patient diagnosis - by gender

SECONDARY OUTCOMES:
Proportion of participants initiated on TPT who completed TPT | Month 18
  Proportion of participants initiated on TPT who completed TPT
Proportion of participants who initiate TPT for whom treatment is discontinued due to adverse events or intolerance in the Intervention phase | Month 18
  Proportion of participants who initiate TPT for whom treatment is discontinued due to adverse events or intolerance in the Intervention phase
Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 4 weeks of the index TB patient diagnosis - overall | Month 18
  Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 4 weeks of the index TB patient diagnosis - overall
Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 4 weeks of the index TB patient diagnosis - by age group (<15, ≥15 years) | Month 18
  Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 4 weeks of the index TB patient diagnosis - by age group (<15, ≥15 years)
Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 4 weeks of the index TB patient diagnosis - by gender | Month 18
  Proportion of HH contacts with newly diagnosed active TB initiated on curative treatment within 4 weeks of the index TB patient diagnosis - by gender

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lienhardt, Study Director — Institut de Recherche pour le Developpement